CLINICAL TRIAL: NCT03586791
Title: Comparison of Pupillometry-guided With Surgical Pleth Index (SPI) Guided General Anesthesia on Perioperative Opioid Consumption and Pain Intensity: a Pilot Study
Brief Title: Comparison of Pupillometry-guided Anesthesia With Surgical Pleth Index Guided Anesthesia
Acronym: PUPIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daegu Catholic University Medical Center (Other)
Responsible Party: Principal Investigator, Eugene Kim, Assistant professor, Daegu Catholic University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: DCMC#5
Record Dates: First submitted 2018-06-30; First posted 2018-07-16 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Cholecystectomy, Laparoscopic; Anesthesia, General; Reflex, Pupillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pupillometry group (Experimental): In this group, anesthesia is performed using Pupillometry guided anesthesia.
  Interventions: Procedure: Pupillometry guided anesthesia
- SPI group (Active Comparator): In this group, anesthesia is performed using SPI guided anesthesia.
  Interventions: Procedure: SPI guided anesthesia
- Control group (Sham Comparator): In this group, remifentanil concentration is controlled by the discretion of the anesthesiologist in charge of the patients (Standard management).
  Interventions: Procedure: Standard management

INTERVENTIONS:
Procedure: Pupillometry guided anesthesia — At least 10 min after anesthesia induction by target-controlled infusion of propofol and remifentanil, baseline values for pupillary diameter is recorded before any surgical procedure.
  During the operation, propofol effect-site target concentration (Ce) is adjusted to maintain the bispectral index (BIS) value between 40 and 60. Remifentanil Ce is adapted every 5 min based on the changes of pupillary diameter. If the pupillary diameter is increased by more than 30% compared to baseline value, remifentanil concentration is increased by 0.5 ng/ml. If the pupillary diameter is maintained between 5 and 30 % change compared with baseline, remifentanil is not modified. In a case of pupillary diameter is decreased less than 5 % change of baseline, remifentanil concentration is decreased by 0.5 ng/ml.
  Other Names: PUPIL
  Arms: Pupillometry group
Procedure: SPI guided anesthesia — During the operation, SPI value should be maintained between 20 and 50 by changing the infusion rate of remifentanil. Even if the SPI is maintained within the target range, the remifentanil infusion rate is increased by 0.5 ng/ml in a case of the SPI value suddenly arises by more than 10.
  Other Names: SPI
  Arms: SPI group
Procedure: Standard management — During the operation, propofol effect-site target concentration (Ce) is adjusted to maintain the bispectral index (BIS) value between 40 and 60.
  Remifentanil concentration is controlled by the discretion of the anesthesiologist in charge of the patients.
  Other Names: Control
  Arms: Control group

SUMMARY:
In this study, the investigators measure a pupil size every 5 minutes during the operation in patients undergoing laparoscopic cholecystectomy under general anesthesia. The investigators would compare the intraoperative opioid consumption and postoperative pain between the group adjusted the anesthetic drug concentration based on the changes of the pupil (Pupil group) and the group based on the changes of a surgical pleth index (SPI group).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20 to 65 yr, American Society of Anesthesiologist Physical status(ASA PS) I to II, scheduled for a laparoscopic cholecystectomy under general anesthesia

Exclusion Criteria:

* Presence of ophthalmologic diseases such as Horner's syndrome or Sjogren's disease.
* Presence of neurologic or metabolic diseases
* Medicated that could interfere with the autonomous nervous system (e.g., b- blockers, anticholinergics)
* History of substance abuse or psychiatric disease
* with chronic pain or preoperative analgesics
* with pacemaker or arrhythmia

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative opioid consumption | During the operation period (Within 2 hour after the anesthesia induction)
  The amount of remifentanil consumption during the operation is calculated by following equation:
  Total remifentanil consumption (mcg) / body weight of the patients (kg)/ duration of anesthesia (min)
Peak pain score assessed by numeric rating scale (NRS) in post-anesthesia care unit (PACU) | During the PACU stay (Within 1 hour after the PACU admission)
  Patients are asked to rate their pain according to the numeric rating scale (NRS, 0=no pain to 10= extreme pain imaginable) every 10 min after the PACU admission. Peak pain score is the peak NRS during PACU stay. Higher NRS represents a worse outcome.

SECONDARY OUTCOMES:
Intraoperative propofol consumption | During the operation period (Within 2 hour after the anesthesia induction)
  The amount of propofol consumption during the operation
Intraoperative vasopressor or vasodilator consumption | During the operation period (Within 2 hour after the anesthesia induction)
  The amount of ephedrine and nicardipine consumption during the operation
PACU stay time | Approximately within 1 hour after the PACU admission
  Duration of time interval from PACU admission to discharge.
Postoperative adverse events | Approximately within 1 hour after the PACU admission
  Check the postoperative nausea and vomiting, dizziness, desaturation, urinary retention, itching sensation and bradycardia
Remnant sedation degree | Approximately within 1 hour after the PACU admission
  Remnant sedation is evaluated by Riker Sedation-Agitation Scale every 10 minutes after the PACU admission.
  1. unarousable, minimal or no response to noxious stimuli, does not communicate of follow commands
  2. very sedate, arouse to physical stimuli but does not communicate or follow command, may move spontaneously
  3. sedate, difficult to arouse but awakens to verbal stimuli or gentle shaking, follows simple commands but drifts off again
  4. Calm and cooperative, calm and follows commands
  5. agitated, anxious or physically agitated and calms to verbal instructions
  6. very agitated, requiring restraint and frequent verbal reminding of limits, biting endotracheal tubes
  7. dangerous agitation, pulling at tracheal tube, trying to remove catheters or striking at staff
Total analgesic consumption after PACU discharge | During 1 day after the operation
  Check the analgesic consumption after PACU discharge including oral, intramuscular and intravenous administration.
Pain score assessed by numeric rating scale (NRS) 1 day after the operation | On 1 day after the operation
  Patients are asked to rate their pain according to the numeric rating scale (NRS, 0=no pain to 10= extreme pain imaginable) 1 day after the operation. Higher NRS represents a worse outcome.
initial Pupillary unrest under ambient light (PUAL) | Just before the induction of anesthesia
  At room light, the pupil is taken for 8 seconds at a frame rate of 30 frames per second. The pupillometer generates raw data in the format of pupil diameter versus time. We define the PUAL as the area under the curve of power spectral density between 0.23 and 3 Hz. The integral of the area is calculated using the composite Simpson's rule.
Pupillary unrest under ambient light (PUAL) on PACU arrival | Approximately within 1 min after the PACU admission
  At room light, the pupil is taken for 8 seconds at a frame rate of 30 frames per second. The pupillometer generates raw data in the format of pupil diameter versus time. We define the PUAL as the area under the curve of power spectral density between 0.23 and 3 Hz. The integral of the area is calculated using the composite Simpson's rule.

OTHER OUTCOMES:
Intraoperative pupil change | Approximately 2 hour after the anesthesia induction
  Measure the pupillary diameter every 5 minutes after the tracheal intubation until the end of operation.
Intraoperative SPI change | Approximately 2 hour after the anesthesia induction
  Check the SPI value throughout the operation using the vital recorder program.
Intraoperative mean blood pressure change | Approximately 2 hour after the anesthesia induction
  Check the mean arterial blood pressure throughout the operation using the vital recorder program.
Intraoperative heart rate change | Approximately 2 hour after the anesthesia induction
  Check the heart rate throughout the operation using the vital recorder program.

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kim, MD, PhD, Study Chair — Assistant professor
Locations (1):
- Eugene Kim, Daegu, Nam-gu, South Korea

REFERENCES:
- [Background] Larson MD, Behrends M. Portable infrared pupillometry: a review. Anesth Analg. 2015 Jun;120(6):1242-53. doi: 10.1213/ANE.0000000000000314. PMID 25988634
- [Background] Huybrechts I, Barvais L, Ducart A, Engelman E, Schmartz D, Koch M. Assessment of thoracic epidural analgesia during general anesthesia using pupillary reflex dilation: a preliminary study. J Cardiothorac Vasc Anesth. 2006 Oct;20(5):664-7. doi: 10.1053/j.jvca.2006.04.004. Epub 2006 Aug 8. PMID 17023285
- [Background] Sabourdin N, Barrois J, Louvet N, Rigouzzo A, Guye ML, Dadure C, Constant I. Pupillometry-guided Intraoperative Remifentanil Administration versus Standard Practice Influences Opioid Use: A Randomized Study. Anesthesiology. 2017 Aug;127(2):284-292. doi: 10.1097/ALN.0000000000001705. PMID 28719527
- [Background] Neice AE, Behrends M, Bokoch MP, Seligman KM, Conrad NM, Larson MD. Prediction of Opioid Analgesic Efficacy by Measurement of Pupillary Unrest. Anesth Analg. 2017 Mar;124(3):915-921. doi: 10.1213/ANE.0000000000001728. PMID 27941575
- [Background] Ledowski T, Burke J, Hruby J. Surgical pleth index: prediction of postoperative pain and influence of arousal. Br J Anaesth. 2016 Sep;117(3):371-4. doi: 10.1093/bja/aew226. PMID 27543532
- [Derived] Kim JH, Jwa EK, Choung Y, Yeon HJ, Kim SY, Kim E. Comparison of Pupillometry With Surgical Pleth Index Monitoring on Perioperative Opioid Consumption and Nociception During Propofol-Remifentanil Anesthesia: A Prospective Randomized Controlled Trial. Anesth Analg. 2020 Nov;131(5):1589-1598. doi: 10.1213/ANE.0000000000004958. PMID 33079883